CLINICAL TRIAL: NCT02173847
Title: Laser Assisted Procedures in Penetrating Keratoplasty: Femtosecond Laser Anvil-shaped Cuts and Laser Welding of the Surgical Wounds
Brief Title: Laser Assisted Procedures in Penetrating Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Santo Stefano (Other)
Collaborators: Istituto di Fisica Applicata (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL-PO-001
Record Dates: First submitted 2014-05-30; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Keratoconus; Corneal Dystrophies; Corneal Opacity
Keywords: anvil-shaped corneal graft; penetrating keratoplasty; femtosecond laser; laser welding
MeSH Terms: conditions — Keratoconus; Corneal Dystrophies, Hereditary; Corneal Opacity | interventions — Keratoplasty, Penetrating; Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Penetrating keratoplasty (Experimental): Femtosecond laser sculptured anvil graft. Diode laser welding of the flap in its final position. 12 months follow up study
  Interventions: Procedure: Penetrating keratoplasty; Device: Femtosecond laser; Device: Diode laser

INTERVENTIONS:
Procedure: Penetrating keratoplasty — Femtosecond laser sculptured anvil graft. Laser welding of the flap in its final position. 12 months follow up study
Device: Femtosecond laser — A commercial femtosecond laser to cut a particular shaped graft
Device: Diode laser — Low power, near infrared diode laser for welding the surgical wound

SUMMARY:
Laser- assisted procedures in penetrating keratoplasty (PK) are proposed to improve the surgical outcomes: minimally invasive procedures, improved biomechanical stability of the transplanted flap, reduction of rejection risks, reduction of inflammation, reduction of infections risk, faster healing process.

In order to achieve these goals, two different lasers were used during PK surgery:

* a femtosecond laser to cut an anvil shaped profile
* a diode laser to weld the surgical wound

DETAILED DESCRIPTION:
The femtosecond laser is used to cut an anvil-shaped laser incision used in PK. This design has the purpose to create a more structurally stable and predictable wound configuration with the aim of a faster recovery of vision and higher optical quality, compared with the conventional blade trephination and the most common laser-cut patterns. The "anvil" profile is designed as described in the followings. Donor and recipient corneal trephination are performed using a 150 kHz FS laser (iFS150TM, IntralaseTM FS Laser, Abbott Medical Optics -AMO, Santa Ana, CA, USA). As concerned iFS150 settings, we refer to the following technical parameters: in the donor graft, the outer and inner diameters of the ring lamellar cut at 350 µm in depth were set at 8.5 mm and 6.6 mm, respectively; the anterior-side cut started with an angle of 135° at a diameter of 7.7 mm, while the straight posterior side cut diameter was 6.7 mm. In the recipient eye, the diameters were designed to be 0.2 mm shorter (8.3 mm outer diameter, 6.4 mm inner diameter, 7.5 mm anterior side cut and 6.5 mm posterior side cut). After completion of the trephination, the corneal button was gently lifted from the host and the donor graft was secured in place on the recipient bed by means of 10-0 nylon cardinal sutures, which were removed after the final 16-running 10-0 nylon suture was completed. A similar FS-laser cut procedure producing a 0.2 mm-narrower corneal bed -diameter is performed on the patient's recipient eye. After completion of the trephination, the corneal button is lifted gently from the host and the donor graft is secured into place with 10-0 nylon cardinal sutures, that are removed as a running 10-0 nylon suture is placed.

The particular "anvil" shape of the graft provides a larger contact surface in between donor and recipient cornea, which enables an effective application of the diode laser welding technique of corneal wounds we have previously set up in cataract and PK applications (Menabuoni et al. 2007, Rossi et al. 2008). This laser-assisted suturing technique is based on the photothermal activation of the stromal collagen, providing an immediate sealing of the surgical wound and a good stabilization of the graft. Once the donor graft was sutured in its final position, diode laser welding was performed. A sterile saturated water solution of 10% w/v Indocyanine Green (ICG) (Pulsion Medical System AG, Munich, Germany) was prepared and applied to the walls of the surgical wound at the donor-recipient interface. A mild photothermal effect was induced by means of a near infrared diode laser (Mod. WELD 800, El.En., Calenzano, FI, Italy) that emitted at 810 nm. The laser light was delivered through a 300-micron core diameter optical fiber that was mounted on a handpiece and used "as a pencil" by the surgeon under a surgical microscope. In a slow, continuous/fluid motion, the surgeon moved the fiber tip along the wound edge at a distance of 1.5 mm from the external surface of the cornea. The power radiation emitted was a 60 mW continuous wave, which resulted in an 8 W/cm2 power density on the tissue surface. The laser welding treatment time was set at 130s.

Thanks two the combine laser assisted procedures, the possible reduction of suture materials allows a faster and improved the healing process, with minimal inflammation and reaction. Thus the combination of FS laser trephination with the diode laser welding technique may provide extremely precise, and minimally invasive surgical procedures in PK.

ELIGIBILITY:
Inclusion Criteria:

* Corneal dystrophy
* keratoconus in its final stages
* post-herpetic leukoma
* corneal scar

Exclusion Criteria:

* systemic diseases
* previous corneal surgery
* glaucoma

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in best spectacle-corrected distance visual acuity (CDVA) | 1 day, 7 days, 1 month, 3 months, 6 months, and 12 months after surgery
  documentation of the visual acuity of patients

SECONDARY OUTCOMES:
Change in objective astigmatism and specular corneal topography | 1 day, 7 days, 1 month, 3 months, 6 months, and 12 months after surgery
  Objective astigmatism and specular corneal topography were evaluated by using a topographer-pachymeter

OTHER OUTCOMES:
Change in anterior segment optical coherence tomography | 1 day, 7 days, 1 month, 3 months, 6 months, and 12 months after surgery
  All patients underwent anterior segment optical coherence tomography to evaluate wound alignment and suture configurations

CONTACTS AND LOCATIONS:
Overall Officials: Luca Menabuoni, MD, Principal Investigator — Head of Corneal and Experimental Surgery at the Department of Ophthalmology
Locations (1):
- U.O. Oculistica Nuovo Ospedale S. Stefano, Prato, Prato, Italy

REFERENCES:
- [Background] Buzzonetti L, Capozzi P, Petrocelli G, Valente P, Petroni S, Menabuoni L, Rossi F, Pini R. Laser welding in penetrating keratoplasty and cataract surgery in pediatric patients: early results. J Cataract Refract Surg. 2013 Dec;39(12):1829-34. doi: 10.1016/j.jcrs.2013.05.046. Epub 2013 Oct 18. PMID 24140371
- [Background] Rossi F, Matteini P, Ratto F, Menabuoni L, Lenzetti I, Pini R. Laser tissue welding in ophthalmic surgery. J Biophotonics. 2008 Sep;1(4):331-42. doi: 10.1002/jbio.200810028. PMID 19343656
- [Background] Menabuoni L, Pini R, Rossi F, Lenzetti I, Yoo SH, Parel JM. Laser-assisted corneal welding in cataract surgery: retrospective study. J Cataract Refract Surg. 2007 Sep;33(9):1608-12. doi: 10.1016/j.jcrs.2007.04.013. PMID 17720078
- [Background] Rossi F, Pini R, Menabuoni L. Experimental and model analysis on the temperature dynamics during diode laser welding of the cornea. J Biomed Opt. 2007 Jan-Feb;12(1):014031. doi: 10.1117/1.2437156. PMID 17343506
- [Background] Rossi F, Pini R, Menabuoni L, Mencucci R, Menchini U, Ambrosini S, Vannelli G. Experimental study on the healing process following laser welding of the cornea. J Biomed Opt. 2005 Mar-Apr;10(2):024004. doi: 10.1117/1.1900703. PMID 15910078
- [Background] Menabuoni L, Canovetti A, Rossi F, Malandrini A, Lenzetti I, Pini R. The 'anvil' profile in femtosecond laser-assisted penetrating keratoplasty. Acta Ophthalmol. 2013 Sep;91(6):e494-5. doi: 10.1111/aos.12144. Epub 2013 Apr 26. No abstract available. PMID 23617376
- [Background] Matteini P, Rossi F, Menabuoni L, Pini R. Microscopic characterization of collagen modifications induced by low-temperature diode-laser welding of corneal tissue. Lasers Surg Med. 2007 Aug;39(7):597-604. doi: 10.1002/lsm.20532. PMID 17868101
- See also: Information about the Ophthalmology Department of the Prato Hospital — http://www.usl4.toscana.it/?act=f&fid=758